CLINICAL TRIAL: NCT05329506
Title: Attitudes and Believes About Vaccinations in a Supportive Care Patient Population
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1070; NCI-2022-00365 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-03-08; First posted 2022-04-15 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-04

CONDITIONS: Vaccinations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Supportive care patient population: Attitudes and Believes About Vaccinations, questionnaires
  Interventions: Other: patient population

INTERVENTIONS:
Other: patient population — questionnaires, standard of care

SUMMARY:
To learn about the attitudes and beliefs towards vaccination both before and after the COVID-19 pandemic in patients who have received supportive care.

DETAILED DESCRIPTION:
Primary Objective:

Our primary objective is to assess patient perception of efficacy and safety of vaccinations.

Secondary Objectives:

To assess demographic predictors of those who would be considered as vaccine hesitant.

To assess patient preferred source of recommendations for or against vaccination.

To assess the role past side effects or allergic reactions play on patient perception of future vaccines.

To assess patient perception of vaccination prior to COVID-19.

To assess patient willingness to get the COVID-19 vaccine.

To assess patient willingness to get the influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are seen as part of a clinic visit with the Supportive Care Clinic at M.D.

   Anderson Cancer Center, also patients who are being seen by the inpatient Supportive Medicine Consultation Service.
2. Patients who are 18 years of age or older
3. Patients who are able to speak English.

Exclusion Criteria:

1. Patients who are unable to sign written consent
2. Patients who are considered delirious at the time of the clinic encounter as defined by a Memorial Delirium Assessment Scale score of 7 or greater. The nursing staff, as a part of the patient intake process and routine care, performs the delirium assessment for clinic patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer Center
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Exploratory survey evaluating the solely patient's opinions and perceptions regarding the safety and efficacy of vaccinations for Parent Attitudes about Childhood Vaccines (PACV-4 scale) with a score of 2 or greater. | through study completion, an average of 1 year
  We will assess the patient's opinion and perception of the safety of vaccinations based upon a questionnaire and a Likert scale of responses.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org